CLINICAL TRIAL: NCT02580747
Title: Clinical Study of Chimeric Mesothelin Antigen Receptor-modified T Cells in Relapsed and/or Chemotherapy Refractory Malignancies
Brief Title: Treatment of Relapsed and/or Chemotherapy Refractory Advanced Malignancies by CART-meso
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, PI, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s2015-080-06
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Malignant Mesothelioma; Pancreatic Cancer; Ovarian Tumor; Triple Negative Breast Cancer; Endometrial Cancer; Other Mesothelin Positive Tumors
MeSH Terms: conditions — Mesothelioma, Malignant; Pancreatic Neoplasms; Ovarian Neoplasms; Triple Negative Breast Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-meso CAR T cells (Experimental): Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  Patients receive anti-meso-CAR retroviral vector-transduced autologous-derived T cells on days 0, 1, 2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: anti-meso-CAR vector transduced T cells

INTERVENTIONS:
Biological: anti-meso-CAR vector transduced T cells — genetically engineered lymphocyte therapy
  Other Names: genetically engineered lymphocyte therapy

SUMMARY:
RATIONALE: Placing a tumor antigen chimeric receptor that has been created in the laboratory into patient autologous or donor-derived T cells may make the body build immune response to kill cancer cells.

PURPOSE: This clinical trial is studying genetically engineered lymphocyte therapy in treating patients with Relapsed and/or Chemotherapy Refractory Advanced Malignancies.

DETAILED DESCRIPTION:
I. Determine the safety and feasibility of the chimeric antigen receptor T cells transduced with the anti-meso vector (referred to as CART-meso cells).

II. Determine duration of in vivo survival of CART-meso cells. RT-PCR (reverse transcription polymerase chain reaction) analysis of whole blood will be used to detect and quantify survival of CART-meso TCR (T-cell receptor) zeta:CD137 over time.

SECONDARY OBJECTIVES:

I. For patients with detectable disease, measure anti-tumor response due to CART-meso cell infusions.

II. Estimate relative trafficking of CART-meso cells to tumor in bone marrow and lymph nodes.

III. For patients with stored or accessible tumor cells determine tumor cell killing by CART-meso cells in vitro.

IV. Determine if cellular or humoral host immunity develops against the murine anti-meso, and assess correlation with loss of detectable CART-meso (loss of engraftment).

V. Determine the relative subsets of CART-meso T cells (Tcm, Tem, and Treg).

ELIGIBILITY:
Inclusion Criteria:

1. Chemotherapy refractory or relapsed mesothelin positive malignant mesothelioma,ovarian tumors,pancreatic cancer,triple negative breast cancer,endometrial cancer and other mesothelin positive tumor
2. Patients must be 18 years of age or older.
3. Patients must have an ECOG (Eastern Cooperative Oncology Group )performance status of 0-2.
4. Patients must have evidence of adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters:

   Absolute neutrophil count greater than 1500/mm3. Platelet count greater than 100,000/mm3. Hemoglobin greater than 10g/dl (patients may receive transfusions to meet this parameter).

   Total bilirubin < 1.5 times upper limits of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m.
5. Seronegative for HIV antibody.
6. Seronegative for active hepatitis B, and seronegative for hepatitis C antibody.
7. Patients must be willing to practice birth control during and for four months following treatment. NOTE: women of child-bearing age must have evidence of negative pregnancy test.
8. Patients must be willing to sign an informed consent.

Exclusion Criteria:

1. Patients with life expectancy less than 12 months will be excluded.
2. Patients with uncontrolled hypertension (> 160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated congestive heart failure (> New York Heart Association Class II), or myocardial infarction within 6 months of study will be excluded.
3. Patients with any of the following pulmonary function abnormalities will be excluded: FEV(forced expiratory volume), < 30% predicted; DLCO (diffusing capacity of lung for carbon monoxide) < 30% predicted (post-bronchodilator); Oxygen Saturation less than 90% on room air.
4. Patients with severe liver and kidney dysfunction or consciousness disorders will be excluded.
5. Pregnant and/or lactating women will be excluded.
6. Patients with active infections, including HIV, will be excluded, due to unknown effects of the vaccine on lymphoid precursors.
7. Patients with any type of primary immunodeficiencies will be excluded from the study.
8. Patients requiring corticosteroids (other than inhaled) will be excluded.
9. Patients with history of T cell tumors will be excluded.
10. Patients who are participating or participated any other clinical trials in latest 30 days will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Study related adverse events | Until week 24
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical

SECONDARY OUTCOMES:
Anti-tumor responses to CART-meso cell infusions | up to 24 weeks

OTHER OUTCOMES:
In vivo existence of CART-meso | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Pediatrics Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China